CLINICAL TRIAL: NCT01941121
Title: CCTG 593: Testing and Linkage to Care, A Multicenter Demonstration Project of the California Collaborative Treatment Group
Brief Title: CCTG 593: Testing and Linkage to Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University of California, Los Angeles (Other); University of Southern California (Other); City of Long Beach Department of Health and Human Services (Other Government); California HIV/AIDS Research Program (Other)
Responsible Party: Principal Investigator, Jill Blumenthal, Associate Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CCTG 593
Record Dates: First submitted 2013-09-09; First posted 2013-09-13 (Estimated); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: HIV Positive; HIV Seronegative
Keywords: HIV Screening; Linkage to PrEP; Linkage to Care; CCTG; 593
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Linkage to PrEP or Care (Experimental): Subjects screened for HIV at any CCTG consortium site will be offered Linkage to PrEP or Care, depending on HIV status. After results are received, HIV testers will obtain verbal consent from the subject to connect with the ALERT Specialist, or otherwise offer the subject the ALERT Specialist contact information. When contacted, the ALERT Specialist will coordinate with the subject the scheduling of the PrEP or Care visit, and remain in contact to ensure linkage.
  Interventions: Behavioral: Linkage to PrEP or Care

INTERVENTIONS:
Behavioral: Linkage to PrEP or Care — Ensuring subjects complete linkage to PrEP or Care through coordinated scheduling and intensive reminders by ALERT Specialist.

SUMMARY:
This is a CCTG sponsored project to determine if those recently screened for HIV would accept assistance to be linked into appropriate health services. After receiving their HIV results, high-risk individuals who test negative will have an option to be linked into a study that offers them Pre-exposure Prophylaxis (PrEP), and individuals who test positive will have an option to be linked into care.

If they accept, tested individuals will be in contact with an ALERT specialist that will help facilitate their linkage. The study's primary analysis will analyze how many HIV screened individuals accept the ALERT specialist assistance.

DETAILED DESCRIPTION:
Design: CCTG 593 is a project to evaluate the uptake and effectiveness of an ALERT specialist serving to

1. link newly diagnosed, HIV infected persons from HIV testing sites to HIV specialist providers, and
2. link confirmed HIV antibody negative persons with continued high risk behaviors to PrEP centers

Duration: Each subject who agrees to linkage will receive ALERT follow-up until successful linkage or 60 days following enrollment for linkage to care or 90 days following enrollment for linkage to PrEP, whichever comes first. The duration of the 593 project will be for 3.5 years or until all subjects have been enrolled and successfully linked, or 60 days pass for linkage to care or 90 days for linkage to PrEP.

Sample Size: Up to 600 subjects will be tested and offered linkage across all CCTG sites: LA County-USC Medical Center, Harbor-UCLA/City of Long Beach Department of Health and Human Services, UCSD/San Diego Health and Human Services Agency.

Study Population: Eligible subjects will include any persons 18 years of age or older who have been tested for HIV at one of the CCTG testing sites (LA County + USC, Long Beach Department of Health and Human Services, and San Diego Health and Human Services Agency).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Has had an HIV test result form the CCTG Consortium testing site as either positive or negative
* Ability to provide informed consent
* English or Spanish Speaking

Exclusion Criteria:

* Severe active substance abuse or mental illness that the investigator feels will interfere with the ability to provide informed consent
* Acute medical illness that requires transfer to a non CCTG hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2013-07-26 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2021-02-09 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects linked to Care or PrEP | Up to 60 days for positives and up to 90 days for negatives from date of HIV screening test
  The primary outcome will measure the proportion of subjects linked a) to HIV care within 60 days of testing HIV-positive or b) to PrEP within 90 days of testing HIV-negative

SECONDARY OUTCOMES:
Acceptance of the linkage program | 60 days from date of HIV screening test
  Secondary outcomes will measure the acceptance of the linkage program, which is defined as those individuals who, after testing either positive or HIV antibody negative, will agree to be contacted by the ALERT specialist.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Jacobson, MD, Study Chair — University of Southern California; Michael Menchine, MD, MPH, Study Chair — University of Southern California; Jill Blumenthal, MD, Principal Investigator — UC San Diego AntiViral Research Center (AVRC)
Locations (3):
- United States (3):
  - City of Long Beach Department of Health and Human Services, Long Beach, California
  - University of Southern California, Los Angeles, California
  - University of California, San Diego, San Diego, California